CLINICAL TRIAL: NCT03829657
Title: A Phase 3, 22-week, Multi-center, Randomized Withdrawal Study of TD-9855 in Treating Symptomatic Neurogenic Orthostatic Hypotension in Subjects With Primary Autonomic Failure
Brief Title: Phase 3 Clinical Effect Durability of TD-9855 for Treating Symptomatic nOH in Subjects With Primary Autonomic Failure
Acronym: REDWOOD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped early due to company decision. Company decision based on analysis results in TD-9855-0169.
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0170; 2018-003941-41 (EudraCT Number)
Record Dates: First submitted 2019-01-10; First posted 2019-02-04 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypotension; MSA; Parkinson's Disease (PD); Pure Autonomic Failure (PAF)
Keywords: Symptomatic Neurogenic Orthostatic Hypotension; symptomatic nOH; multiple symptom atrophy; MSA; Parkinson's disease; PD; pure autonomic failure; PAF; orthostatic hypotension; OH; REDWOOD; ampreloxetine; low blood pressure; dizziness; fainting; blacking out; lightheadedness; norepinephrine; hypotension; Neurogenic Orthostatic Hypotension; nOH; 170; 0170; 145; 0145; TD-9855; TD9855; Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Pure Autonomic Failure; Hypotension, Orthostatic; Hypotension; Dizziness; Syncope; Parkinsonian Disorders | interventions — ampreloxetine

STUDY DESIGN:
Intervention Model Description: Open Label Extension followed by Randomized Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ampreloxetine (Open Label (OL)) (Experimental): Participants will receive ampreloxetine as a single, oral, daily dose of active drug for 16 weeks.
  Interventions: Drug: ampreloxetine
- ampreloxetine (Experimental): After completing the OL, participants randomized to ampreloxetine will receive single, oral, daily dose of active drug for a further 6 weeks.
  Interventions: Drug: ampreloxetine
- Placebo (Placebo Comparator): After completing the OL, participants randomized to Placebo will receive single, oral, daily dose of placebo for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ampreloxetine — Oral tablet, QD (Daily)
  Other Names: TD-9855
  Arms: ampreloxetine; ampreloxetine (Open Label (OL))
Drug: Placebo — Oral tablet, QD
  Arms: Placebo

SUMMARY:
A Phase 3, 22-week, Multi-center, Randomized Withdrawal Study of ampreloxetine in Treating Symptomatic Neurogenic Orthostatic Hypotension in Subjects with Primary Autonomic Failure

DETAILED DESCRIPTION:
Phase 3, multi-center, randomized withdrawal study to evaluate the sustained benefit in efficacy and safety of ampreloxetine in subjects with primary autonomic failures (MSA, PD, or PAF) and symptomatic nOH. The study consists of 3 periods: (i) 16-week open-label (OL) treatment with ampreloxetine, (ii) 6-week randomized placebo-controlled treatment, and (iii) 2-week follow-up (only for patients who do not enroll in Study 0171 (long-term extension safety study)).

ELIGIBILITY:
Inclusion Criteria (For 0169 Completers Group):

* Subject has completed 4 weeks of double blind treatment in Study 0169 (V6) and, in the opinion of the Investigator, could benefit from continued treatment with ampreloxetine. Only subjects with OHSA#1 score of ≤7 will be eligible for randomization for the double-blind treatment period.
* Subject has a minimum of 80% study medication compliance in Study 0169.

Inclusion Criteria (For De Novo Group):

* Subject is male or female and at least 30 years old.
* Subject must meet the diagnostic criteria of symptomatic nOH, as demonstrated by a sustained reduction in BP of ≥20 mm Hg (systolic) or ≥10 mm Hg (diastolic) within 3 min of being tilted-up ≥60o from a supine position as determined by a tilt-table test.
* Subject must score at least a 4 on the OHSA#1 at V1.
* For subjects with PD only: Subject has a diagnosis of PD according to the United Kingdom Parkinson's Disease Society (UKPDS) Brain Bank Criteria (1992).
* For subjects with MSA only: Subject has a diagnosis of possible or probable MSA of the Parkinsonian subtype (MSA-P) or cerebellar subtype (MSA-C) according to The Gilman Criteria (2008).
* For subjects with PAF only: Subject has documented impaired autonomic reflexes, including the Valsalva maneuver performed within 24 months from the date of randomization
* Subject has plasma Norepinephrine (NE) levels ≥ 100 pg/mL after being in seated position for 30 minutes.

Exclusion Criteria (For 0169 Completers Group):

* Subject has a medical, laboratory, or surgical issue(s) deemed by the investigator to be clinically significant.
* Subject has an uncooperative attitude or reasonable likelihood of non-compliance with the protocol.
* Subject has a concurrent disease or condition that, in the opinion of the investigator, would confound or interfere with study participation or evaluation of safety, tolerability, or pharmacokinetics of the study drug.

Exclusion Criteria (For De Novo Group):

* Subject has a known systemic illness known to produce autonomic neuropathy, including but not limited to amyloidosis, and autoimmune neuropathies.
* Subject has a known intolerance to other NRIs or serotonin norepinephrine reuptake inhibitors (SNRIs).
* Subject currently uses concomitant antihypertensive medication for the treatment of essential hypertension unrelated to autonomic dysfunction.
* Subject has used strong CYP1A2 inhibitors or inducers within 7 days or 5 half-lives, whichever is longer, prior to V1 or requires concomitant use until the follow-up visit.
* Subject has changed dose, frequency, or type of prescribed medication for orthostatic hypotension within 7 days prior to V1.

  * Midodrine and droxidopa (if applicable) must be tapered off at least 7 days prior to V1.
* Subject has known or suspected alcohol or substance abuse within the past 12 months (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision [DSM-IV-TR®] definition of alcohol or substance abuse).
* Subject has a clinically unstable coronary artery disease, or has had a major cardiovascular or neurological event in the past 6 months.
* Subject has used any monoamine oxidase inhibitor (MAO-I) within 14 days prior to V1.
* Subject has a history of untreated closed angle glaucoma, or treated closed angle glaucoma that, in the opinion of an ophthalmologist, might result in an increased risk to the subject.
* Subject has any significant uncontrolled cardiac arrhythmia.
* Subject has a Montreal Cognitive Assessment (MoCA) ≤23.
* Subject is unable or unwilling to complete all protocol specified procedures including questionnaires.
* Subject had a myocardial infarction in the past 6 months or has current unstable angina.
* Subject has known congestive heart failure (New York Heart Association [NYHA] Class 3 or 4).
* Subject has a clinically significant abnormal laboratory finding (e.g., alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >3.0 x upper limit of normal [ULN]; blood bilirubin [total] >1.5 x ULN; estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2, or any abnormal laboratory value that could interfere with safety of the subject).
* Subject has demonstrated a history of lifetime suicidal ideation and/or suicidal behavior, as outlined by the Columbia Suicide Severity Rating Scale (C-SSRS)(Baseline/Screening Version). Subject should be assessed by the rater for risk of suicide and the subject's appropriateness for inclusion in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (82):
- United States (20):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - UC San Diego Movement Disorder Center, La Jolla, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Colorado Springs Neurological Associates, PC, Colorado Springs, Colorado
  - Parkinson's Disease and Movement Disorders Center, Boca Raton, Florida
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Neurostudies, Inc, Port Charlotte, Florida
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University Health System, Glenview, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - New York University Langone Health, New York, New York
  - Wake Forest University Baptist Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center (UCGNI), Cincinnati, Ohio
  - Ohio State University - Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Georgetown University Hospital, McLean, Virginia
  - Inland Northwest Research, Spokane, Washington
- Australia (4):
  - Concord Hospital, Neurosciences Department, Concord, New South Wales
  - Clinical Trials Centre, Level 3 Monash Health Translational Precinct Building Monash Medical Centre, Clayton, Victoria
  - The Royal Melbourne Hospital Neurology Department, Parkville, Victoria
  - Perron Institute for Neurological and Translational Science, Nedlands, Western Australia
- Austria (2):
  - Medizinische Universitat Innsbruck, Abteilung fur Neurologie, Innsbruck
  - Universitatsklinikum Tulln Abteilung fur Neurologie, Tulln
- MHATNP Sv. Naum EAD Clinic of Neurological Diseases for Locomotor Disorders, Sofia, Bulgaria
- Canada (3):
  - University of Calgary Teaching Research and Wellness Building, Calgary, Alberta
  - Toronto Western Hospital, Toronto, Ontario
  - Montreal Neurological Institute & Hospital, Montreal, Quebec
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Odense Universitetshospital, Odense
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - Astra Team Clinic, Tallinn
  - Tartu University Hospital, Tartu
- CHU de Nîmes - Hôpital Caremeau, Nîmes, France
- Germany (3):
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Charite - Campus Virchow-Klinikum, Klinik fur Neurologie, Berlin
  - Praxis Dr. med. Christian Oehlwein, Gera
- Semmelweis Egyetem, Neurologiai Klinika, Budapest, Hungary
- Israel (3):
  - Rabin Medical Center, Beilinson Campus, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Universita di Bologna-Clinica Neurologica - Dipt di Scienze Neurologiche Ospedale Bellaria, Bologna
  - Azienda Ospedaliera Universitaria Policlinico - Vittorio Emanuele (Presidio Gaspare Rodolico), Catania
  - Universita degli studi Gabriele D' Annunzio Chieti, Chieti
  - Fondazione IRCCS CA Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero-Universitaria Pisana- Ospedale S. Chiara, U.O. di Neurologia - Neurofisiopatologia, Pisa
  - Fondazione PTV - Policlinico Tor Vergata I U.0.C. Neurologia, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS / Istituto di Neurologia - Ambulatorio Disturbi del Movimento, Roma
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - A.O. Santa Maria, Terni
- New Zealand Brain Research Institute, Christchurch, New Zealand
- Poland (6):
  - Specjalistyczna Praktyka Lekarska, Prof. Grzegorz Opala, Katowice
  - Krakowska Akademia Neurologii Sp. Zo.o. Centrum Neurologii Klinicznej, Krakow
  - Instytut Zdrowia dr Boczarska-Jedynak, Oświęcim
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Siemianowice Śląskie
  - ETG Warszawa, Warsaw
  - Specjalistyczne Gabinety sp. z o.o., Warsaw
- Portugal (2):
  - Hospital da Senhora da Oliveira Guimarães, Guimarães
  - CNS-Campus Neurologico Senior, Torres Vedras
- Russia (6):
  - Saint Petersburg State Budgetary Institution of Healthcare City Hospital #40 of Kurortnyi Region, Saint Petersburg, Sestroretsk
  - FSBI Federal Sibirian Scientific and Clinical Center of Federal Medico-Biological Agency, Krasnoyarsk
  - State Budgetary Institution of Healthcare of Novosibirsk region City Clinical Hospital #34, Novosibirsk
  - City Neurological Center Sibneiromed, LLC, Novosibirsk
  - FSBI National Medical Research Centre of psychiatry and neurology named after V.M. Bekhterev of the MOH of the Russian Federation, Saint Petersburg
  - FSBI of Science Institute of Human Brain named after N .P. Bekhtereva of Russian Academy of Sciences, Saint Petersburg
- Spain (5):
  - Hospital Universitario Mutua de Terrasa, Terrassa, Barcelona
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital de Cruces, Bilbao, Vizcaya
  - Hospital del Mar, Barcelona
  - Hospital Universitario de La Princesa, Madrid
- Ukraine (3):
  - Communal Noncommercial Enterprise City Policlinic #9 of Kharkiv City Council, Kharkiv
  - Communal Noncommercial Enterprise of Lviv Regional Council Lviv Regional Clinical Hospital, Lviv
  - Communal Institution Acad. O.I. Yuschenko VRPsH Vinnytsia M.I. Pyrogov NMU Ch of ND with the Course of Neurosurgery, Vinnytsia
- United Kingdom (7):
  - Royal Devon and Exeter Hospital NHS Trust, Exeter, Devon
  - Cognition Health Unit 2, Plymouth, Devon
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - Clinical Research Centre, William Harvey Heart Centre, London
  - King's College Hospital, London
  - Re:Cognition Health Ltd, London
  - The National Hospital for Neurology & Neurosurgery, London

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from February 2019 to November 2021. 203 participants were enrolled in the open label (OL) treatment period, including 170 participants from the 0169 study (NCT number: NCT03750552). 128 participants who completed the OL treatment period continued in the randomized withdrawal (RW) treatment period.
Groups:
- OL Treatment Period: 0169 Placebo Rollover: Participants who received the placebo in study 0169, received 10 mg oral ampreloxetine once a day (QD) for up to 16 weeks.
- OL Treatment Period: 0169 Ampreloxetine Rollover: Participants who received ampreloxetine in study 0169, received 10 mg oral ampreloxetine QD for up to 16 weeks.
- OL Treatment Period: De Novo: Participants with symptomatic neurogenic orthostatic hypotension (nOH) who met all applicable study inclusion criteria and none of the applicable exclusion criteria, received 10 mg oral ampreloxetine QD for up to 16 weeks. These participants did not roll over from the 0169 study.
- RW Treatment Period: Placebo: Participants who completed the OL treatment period and were randomized to receive oral placebo QD for a further 6 weeks in the RW treatment period.
- RW Treatment Period: Ampreloxetine: Participants who completed the OL treatment period and were randomized to receive 10 mg oral ampreloxetine QD for a further 6 weeks in the RW treatment period.
Period: OL Treatment Period (Week 1 to Week 16)
Arm/Group | OL Treatment Period: 0169 Placebo Rollover | OL Treatment Period: 0169 Ampreloxetine Rollover | OL Treatment Period: De Novo | RW Treatment Period: Placebo | RW Treatment Period: Ampreloxetine
Started | 85 | 85 | 33 | 0 | 0
Completed | 52 | 64 | 12 | 0 | 0
Not Completed | 33 | 21 | 21 | 0 | 0
Not completed — Adverse Event | 12 | 4 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 3 | 9 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 7 | 5 | 0 | 0
Not completed — Failure to Meet Day 29 Continuation Criterion | 10 | 6 | 4 | 0 | 0
Not completed — Miscellaneous | 3 | 1 | 1 | 0 | 0
Period: RW Treatment Period (Week 16 to Week 24)
Arm/Group | OL Treatment Period: 0169 Placebo Rollover | OL Treatment Period: 0169 Ampreloxetine Rollover | OL Treatment Period: De Novo | RW Treatment Period: Placebo | RW Treatment Period: Ampreloxetine
Started | 0 | 0 | 0 | 64 | 64
Completed | 0 | 0 | 0 | 61 | 58
Not Completed | 0 | 0 | 0 | 3 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: OL Treatment Period Safety Analysis Set: all enrolled participants who received at least 1 dose of ampreloxetine during the OL period.
Groups:
- Total: Total of all reporting groups
Arm/Group | OL Treatment Period: 0169 Placebo Rollover | OL Treatment Period: 0169 Ampreloxetine Rollover | OL Treatment Period: De Novo | Total
Number analyzed (Participants) | 83 | 85 | 32 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (9.35) | 68.2 (9.00) | 69.0 (7.97) | 68.4 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 8 | 60
  Male | 61 | 55 | 24 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 0 | 6
  Not Hispanic or Latino | 77 | 76 | 32 | 185
  Unknown or Not Reported | 4 | 5 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 80 | 83 | 31 | 194
  Black or African American | 0 | 1 | 1 | 2
  Asian | 2 | 1 | 0 | 3
  Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Treatment Failure at Week 6 of RW Treatment Period
Description: Treatment failure was defined as proportion of participants who met the following criteria at Week 6 following randomization: Change (worsening) from baseline in Question 1 of the Orthostatic Hypotension Symptom Assessment (OHSA#1) score of 1.0 point and worsening of disease severity as assessed by a 1-point change in Patient Global Impression of Severity (PGI-S). OHSA Question #1 assessed dizziness, lightheadedness, feeling faint, or feeling like you might blackout. PGI-S assessed patient's impression of disease severity.
  Least squares mean here is the model-based proportion of participants with treatment failure using logistic regression.
Time Frame: 6-week randomized withdrawal period (Week 16 to Week 22)
Population: RW Treatment Period Full Analysis Set: all randomized participants who received at least 1 dose of study medication (ampreloxetine or placebo) following randomization.
Measure: Least Squares Mean (Standard Error); unit: Proportion of participants
Arm/Group | RW Treatment Period: Placebo | RW Treatment Period: Ampreloxetine
Number analyzed (Participants) | 64 | 64
Proportion of participants | 0.42 (0.068) | 0.30 (0.065)
Statistical Analysis 1: Comparison: RW Treatment Period: Placebo vs RW Treatment Period: Ampreloxetine; Test type: Superiority; p = 0.196, Regression, Logistic; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.27 to 1.29]

ADVERSE EVENTS:
Time Frame: OL Treatment Period: Day 1 to Week 16 (plus a 2 week follow-up period); RW Treatment Period: Week 16 to Week 24 (plus a 2 week follow-up period)
Description: OL Safety Analysis Set: all enrolled participants who received at least 1 dose of ampreloxetine during the OL period.
  RW Treatment Safety Analysis Set: all randomized participants who received at least 1 dose of study medication (ampreloxetine or placebo) following randomization. The Safety Analysis Set and FAS were identical for the RW treatment period.
Arm/Group | OL Treatment Period: 0169 Placebo Rollover | OL Treatment Period: 0169 Ampreloxetine Rollover | OL Treatment Period: De Novo | RW Treatment Period: Placebo | RW Treatment Period: Ampreloxetine
All-Cause Mortality (participants affected / at risk) | 2/83 | 3/85 | 0/32 | 0/64 | 2/64
Serious Adverse Events (participants affected / at risk) | 7/83 | 8/85 | 1/32 | 2/64 | 4/64
Other Adverse Events (participants affected / at risk) | 41/83 | 48/85 | 16/32 | 16/64 | 17/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OL Treatment Period: 0169 Placebo Rollover (N=83) | OL Treatment Period: 0169 Ampreloxetine Rollover (N=85) | OL Treatment Period: De Novo (N=32) | RW Treatment Period: Placebo (N=64) | RW Treatment Period: Ampreloxetine (N=64)
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bulbar palsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Subcapsular renal haematoma (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OL Treatment Period: 0169 Placebo Rollover (N=83) | OL Treatment Period: 0169 Ampreloxetine Rollover (N=85) | OL Treatment Period: De Novo (N=32) | RW Treatment Period: Placebo (N=64) | RW Treatment Period: Ampreloxetine (N=64)
Urinary tract infection (Infections and infestations) | 2 | 8 | 2 | 3 | 2
Headache (Nervous system disorders) | 5 | 3 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 4 | 3 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 5 | 2 | 0 | 0
Syncope (Nervous system disorders) | 2 | 2 | 0 | 0 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
On and off phenomenon (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness exertional (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypokinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Multiple system atrophy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Oromandibular dystonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Radial nerve palsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Spasmodic dysphonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Bruxism (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Hypomania (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hair growth rate abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0
Colonoscopy (Investigations) | 0 | 0 | 1 | 0 | 0
Glomerular filtration rate abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Supine hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
White coat hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Open angle glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Allergy to vaccine (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Priapism (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Device occlusion (Product Issues) | 0 | 1 | 0 | 0 | 0
Walking disability (Social circumstances) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cystoscopy (Investigations) | 0 | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Uterine enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Bulbar palsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
De Novo participants in the OL treatment period had limited follow-up due to early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT03829657/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT03829657/SAP_001.pdf